CLINICAL TRIAL: NCT06394739
Title: RevCore for In Stent Thrombosis (REVIT)
Brief Title: RevCore for In Stent Thrombosis
Acronym: REVIT
Status: Recruiting | Type: Observational
Sponsor: Inari Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 23-002 REVIT
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-02

CONDITIONS: In-stent Thrombosis
MeSH Terms: interventions — Thrombectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Thrombectomy — RevCore Thrombectomy to treat in-stent thrombosis
  Other Names: RevCore Thrombectomy

SUMMARY:
The purpose of this research is to collect information about how the RevCore Thrombectomy Catheter works to treat stent blockages.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients with stent age > 6 weeks
3. Location of thrombosed stents in proximal lower extremity deep vein segments including at least common femoral, external iliac, or common iliac vein
4. RevCore Thrombectomy Catheter must enter vasculature
5. Willing and able to provide informed consent

Exclusion Criteria:

1. Exposed stents with broken struts, significantly deformed struts, struts protruding into the vessel
2. Stents not wall apposed
3. Stents compressed to <10mm
4. Bilateral in-stent thrombosis
5. Congenital anatomic anomalies of the iliac veins
6. Allergy, hypersensitivity, or thrombocytopenia from heparin or iodinated contrast agents, except for mild to moderate contrast allergies for which pretreatment can be used
7. Any contraindication to anticoagulants or antiplatelets that, in the opinion of the Investigator, cannot be medically managed throughout the study period
8. Chronic non-ambulatory status
9. Known hypercoagulable states (e.g. antiphospholipid syndrome) that, in the opinion of the Investigator, cannot be medically managed throughout the study period
10. Inability to secure venous access
11. Subject has any condition for which, in the opinion of the Investigator, participation would not be in the best interest of the subject
12. Current participation in another investigational drug or device treatment study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 100 subjects with in-stent thrombosis will be enrolled. All subjects who sign informed consent and who meet all of the inclusion criteria and none of the exclusion criteria will be eligible to participate in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Evidence of successful stent recanalization | Immediately after the RevCore thrombectomy procedure for in-stent thrombosis
  Defined as patency ≥50% luminal diameter utilizing intravascular ultrasound (IVUS)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Yale University, New Haven, Connecticut
  - Medstar Health Research Institute, Washington D.C., District of Columbia
  - University of Maryland, Baltimore, Maryland
  - New York University- Langone, New York, New York
  - Mission Health, Asheville, North Carolina
  - UH Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny Health Network Research Institute, Pittsburgh, Pennsylvania
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - El Paso Cardiology Associates, El Paso, Texas
  - Sentara, Norfolk, Virginia
  - University of Washington, Seattle, Washington
  - West Virginia University- Ruby Memorial, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Undecided